CLINICAL TRIAL: NCT03312790
Title: Effects of Augmented Reality Glasses on Muscle Activity, Balance, Physical and Mental Fatigue
Brief Title: Effects of Augmented Reality on Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Burgundy (Other)
Responsible Party: Principal Investigator, Nicolas Babault, principal investigator, University of Burgundy
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: CEP1701
Record Dates: First submitted 2017-06-13; First posted 2017-10-18 (Actual); Last update posted 2017-10-18 (Actual); Status verified 2017-10

CONDITIONS: Physical Activity; Mental Status Change
Keywords: augmented reality; fatigue; muscle; heart rate; mental function
MeSH Terms: conditions — Motor Activity; Fatigue

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- augmented reality device (Experimental): Tasks realized using augmented reality device
  Interventions: Device: Tasks
- Real condition (Other): Same tasks than augmented reality realized in normal/real condition
  Interventions: Device: Tasks

INTERVENTIONS:
Device: Tasks — Augmented reality device Real condition
  Other Names: Workers tasks

SUMMARY:
Nowadays, augmented reality (AR) has gained attention but little is known concerning its repercussion in individuals when considering some mental and physiological aspects. Therefore, the aim of this study was to investigate the effects of AR glasses on some cognitive and physiological functions in an attempt to determine its safety for workers.

DETAILED DESCRIPTION:
Twelve volunteers were tested during two separate randomized sessions: one with AR glasses (ARGlass) and one in normal condition (Normal). Participants had two perform different tasks of a 90 minutes total duration. Before, during and after these tasks, two feet balance, one foot balance, precision balance, stroop and memory tests were performed. Also, heart rate and electromyographic activity of some muscles were recorded. Finally a survey was filled to determine, for example fatigue, pain or comfort.

ELIGIBILITY:
Inclusion Criteria:

* healthy
* BMI < 27
* physically active
* informed consent written form

Exclusion Criteria:

* in-habitual fatigue
* taking drugs and alcohol more than twice a day
* potential psychomotor disease
* injury in the preceding 3 months
* no healthcare

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-02-15 (Actual); Study Completion 2017-03-01 (Actual)

PRIMARY OUTCOMES:
Voluntary activation using electromyography of upper and lower limb muscles | Measured just before and immediately after every 30 minutes series (repeated three times)
  The mean electromyographic activity of trapezius, deltoideus, biceps brachii, latissimus dorsi, soleus and tibialis anterior muscles will be measured using surface electrodes

SECONDARY OUTCOMES:
Heart rate | Measured just before and immediately after every 30 minutes series (repeated three times)
  Heart rate during the different tasks and test session
Balance | Measured just before and immediately after every 30 minutes series (repeated three times)
  Two feet, one foot and precision tasks balance (center of pressure displacement)
Memory | Measured just before and immediately after every 30 minutes series (repeated three times)
  5 words memory test
attention | Measured just before and immediately after every 30 minutes series (repeated three times)
  Stroop test
subjective perceived exertion | Measured just before and immediately after every 30 minutes series (repeated three times)
  difficulty of the tasks using a visual analogic scale
subjective pain perception | Measured just before and immediately after every 30 minutes series (repeated three times)
  pain perceived (visual analogic scale) and the location if some pain sensation
subjective fatigue perception | Measured just before and immediately after every 30 minutes series (repeated three times)
  perceived fatigue (visual analogic scale) and the location in case of fatigue feeling

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Babault, PhD, Principal Investigator — University of Burgundy
Locations (1):
- Centre d'Expertise de la Performance - Université de Bourgogne, Dijon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Babault N, Paizis C, Deley G, Guerin-Deremaux L, Saniez MH, Lefranc-Millot C, Allaert FA. Pea proteins oral supplementation promotes muscle thickness gains during resistance training: a double-blind, randomized, Placebo-controlled clinical trial vs. Whey protein. J Int Soc Sports Nutr. 2015 Jan 21;12(1):3. doi: 10.1186/s12970-014-0064-5. eCollection 2015. PMID 25628520
- See also: centre d'expertise de la performance — http://www.cepcometti.com